CLINICAL TRIAL: NCT07057388
Title: Comparison of Postoperative Pain Using Two Different Obturation Techniques: Single Cone Versus Continuous Wave Compaction
Brief Title: Postoperative Pain: Single Cone vs Continuous Wave Compaction Obturation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Principal Investigator, Samia Rasool, post graduate resident, CMH Lahore Medical College and Institute of Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107/CIV/Trg/Op/16/24
Record Dates: First submitted 2025-06-20; First posted 2025-07-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-01

CONDITIONS: Root Canal Obturation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group one receiving cold lateral condensation obturation (No Intervention): conventional method of obturation is used
- Group 2 receiving obturation through continous wave compaction (Experimental): heated gutta percha using continous wave compaction
  Interventions: Device: continous wave compaction

INTERVENTIONS:
Device: continous wave compaction — post operative pain measurement using continous wave compaction
  Arms: Group 2 receiving obturation through continous wave compaction

SUMMARY:
The study involves two groups in which root canal obturation will be performed using different obturation techniques. Group one consists of participants with the single cone cold lateral condensation method, while group two consists of participants with the continuous wave compaction technique. Postoperative pain will be assessed and compared between the two groups.

DETAILED DESCRIPTION:
This study aims to compare postoperative pain levels following root canal obturation using two different techniques: the single cone cold lateral condensation method and the continuous wave compaction technique. Participants will be divided into two groups, each receiving one of the two obturation methods. Pain levels will be evaluated at defined preoperative and postoperative intervals to determine if there is a significant difference in patient-reported outcomes between the techniques. The findings may contribute to clinical decision-making regarding the selection of obturation methods to minimize patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* irreversible pulpitis

Exclusion Criteria:

* periapical abcess

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
comparison of post operative pain | 24 hours , 48 hours and 1week
  post operative pain using VISUAL ANALOGUE SCALE (VAS) , two methods of obturation to assess pain after root canal using cold lateral versus heated gutta percha Pre operative pain will be measured on each patient according to visual analogue scale as baseline before intiating the procedure .

CONTACTS AND LOCATIONS:
Overall Officials: Imran Khan, BDS FCPS, Study Director — 28 military dental centre
Locations (1):
- 28 Military Dental Centre, Lahore, Punjab Province, Pakistan